CLINICAL TRIAL: NCT00620750
Title: Extended-release Naltrexone (Vivitrol) for the Treatment of Alcohol Dependence in Urban Primary Care: a Feasibility Study
Brief Title: Extended-release Naltrexone for Alcohol Dependence in Primary Care
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Alkermes, Inc. (Industry)
Responsible Party: Principal Investigator, Marc Gourevitch, Director of General Internal Medicine, NYU Langone Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C18816/6067/DP/US
Record Dates: First submitted 2008-02-11; First posted 2008-02-21 (Estimated); Results first posted 2011-09-27 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2011-08

CONDITIONS: Alcohol Dependence
Keywords: Alcohol dependence
MeSH Terms: conditions — Alcoholism | interventions — vivitrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Extended release injectable naltrexone (Experimental)
  Interventions: Drug: Extended release injectable naltrexone (Vivitrol)

INTERVENTIONS:
Drug: Extended release injectable naltrexone (Vivitrol) — Three sequential monthly injections of extended release injectable naltrexone (Vivitrol), with option to extend participation for an additional 12 months.
  Other Names: Vivitrol

SUMMARY:
Naltrexone is an opioid antagonist with a high affinity for the mu opioid receptor. The efficacy of extended-release naltrexone (Vivitrol) as a treatment for alcohol dependence has been demonstrated in clinical trials, raising the prospect of integrating pharmacologic treatment for alcohol dependence into general medical care settings. However, the feasibility of implementing this United States Food and Drug Administration approved treatment in the front-line settings in which it is most needed has not been demonstrated. This is an open-label pilot feasibility study of implementing treatment with Vivitrol in primary care medical clinics in a safety net hospital system affiliated with an urban academic center.

ELIGIBILITY:
Inclusion Criteria:

* Current alcohol dependence
* Age 18 or older
* English or Spanish-speaking
* Without untreated severe mental illness
* Liver enzymes (alanine aminotransferase and aspartate aminotransferase) ≤ 3x normal
* Kept 2 of last 3 clinic primary care appointments and/or has a working telephone number at which can be contacted directly
* Either a) currently abstinent (e.g., referred from an inpatient 'detox' setting) or b) with the ability, in the clinician's judgment, to achieve and maintain abstinence
* If female of child-bearing potential, must be using adequate contraception
* Able to understand study procedures

Exclusion Criteria:

* Currently opioid dependent or requiring ongoing treatment with opioids for any indication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2007-07; Primary Completion 2008-11 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc N Gourevitch, MD, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU School of Medicine, New York, New York, United States

REFERENCES:
- [Result] Lee JD, Grossman E, DiRocco D, Truncali A, Hanley K, Stevens D, Rotrosen J, Gourevitch MN. Extended-release naltrexone for treatment of alcohol dependence in primary care. J Subst Abuse Treat. 2010 Jul;39(1):14-21. doi: 10.1016/j.jsat.2010.03.005. Epub 2010 Apr 2. PMID 20363090
- [Derived] Lee JD, Grossman E, Huben L, Manseau M, McNeely J, Rotrosen J, Stevens D, Gourevitch MN. Extended-release naltrexone plus medical management alcohol treatment in primary care: findings at 15 months. J Subst Abuse Treat. 2012 Dec;43(4):458-62. doi: 10.1016/j.jsat.2012.08.012. Epub 2012 Sep 15. PMID 22985676

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study began July 2007. Community recruitment was performed from August 2007 to September 2008 in the primary care clinics of Bellevue Hospital and Gouverneur Diagnostic and Treatment Centers, two public hospital facilities in lower Manhattan. 116 persons contacted study staff regarding possible participation, and 76 were consented and screened.
Pre-assignment Details: Four consented patients were ineligible due to elevated liver function tests (n = 2), opioid dependence (n =1), and an uncontrolled psychiatric condition (n = 1). Seventy two participants met eligibility criteria and consented to study involvement, sixty-five participants presented for the initial treatment visit.
Groups:
- Extended Release Injectable Naltrexone: This was a single arm trial, with no formal control group. The treatment administered was a single 380-mg extended-release naltrexone (Vivitrol)dose injected intramuscularly into the upper, outer gluteus,alternating sides monthly. Medication injection was performed by physicians per package insert guidelines. A final Month 4 visit assessed treatment outcomes and satisfaction. Patients interested in further extended-release naltrexone treatment at study end were referred to a related 12-month extended-release naltrexone extension study, and all patients were able to continue in primary care.
Period: Overall Study
Arm/Group | Extended Release Injectable Naltrexone
Started | 65
Completed | 40
Not Completed | 25
Not completed — Lost to Follow-up | 25

BASELINE CHARACTERISTICS:
Arm/Group | Extended Release Injectable Naltrexone
Number analyzed (Participants) | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 65
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 46 (8.535196)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 49
Region of Enrollment [Number; unit: participants]
  United States | 65

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients Initiating Vivitrol Treatment Who Receive 3 Consecutive Monthly Vivitrol Injections
Time Frame: 4 months
Population: Per protocol
Measure: Number; unit: Percent of participants
Arm/Group | Extended Release Injectable Naltrexone
Number analyzed (Participants) | 65
Percent of participants | 40

ADVERSE EVENTS:
Arm/Group | Extended Release Injectable Naltrexone
Serious Adverse Events (participants affected / at risk) | 2/65
Other Adverse Events (participants affected / at risk) | 45/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Extended Release Injectable Naltrexone (N=65)
Severe injection site reaction (Injury, poisoning and procedural complications) | 1 (1)
unexpected pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Extended Release Injectable Naltrexone (N=65)
any injection site reaction (Injury, poisoning and procedural complications) | 30 (30)
nausea (Gastrointestinal disorders) | 18 (18)
fatigue (General disorders) | 8 (8)
headache (General disorders) | 6 (6)
flu-like symptoms (General disorders) | 6 (6)
insomnia (General disorders) | 6 (6)
AST/ALT >5x normal (General disorders) | 2 (2)
other complaints (General disorders) | 22 (22)

LIMITATIONS AND CAVEATS:
There was no formal control arm. Drinking and satisfaction outcomes were self-reported, these outcomes and Adverse Event data were not available for those lost to follow-up. The drinking Timeline Follow-Back is subject to recall and response biases.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No